CLINICAL TRIAL: NCT02355782
Title: Provision of OMS721 to Patients With Thrombotic Microangiopathy Under Compassionate Use
Brief Title: OMS721 Compassionate Use in Patients With Thrombotic Microangiopathy
Status: Available | Type: Expanded Access
Sponsor: Michal Nowicki (Other)
Responsible Party: Sponsor-Investigator, Michal Nowicki, Professor, Medical University of Lodz
Organization: Medical University of Lodz (Other)
Other Study IDs: TMA-100
Record Dates: First submitted 2015-01-28; First posted 2015-02-04 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-01

CONDITIONS: Thrombotic Microangiopathy
Keywords: TMA, aHUS, TTP, stem cell transplant-associated TMA
MeSH Terms: conditions — Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome | interventions — narsoplimab

INTERVENTIONS:
Biological: OMS721 — Human IgG4 MASP-2 Monoclonal Antibody

SUMMARY:
The purpose of this compassionate use study, for two patients with thrombotic microangiopathy, is to provide expanded access to patients who have participated in the clinical trial OMS721-TMA-001 and in whom improvement in their disease markers was observed while on treatment or to patients who could otherwise benefit from the treatment. This is a treatment protocol; not a research protocol.Therefore, only patients in study OMS721-TMA-001 deemed eligible by the investigator may participate.

DETAILED DESCRIPTION:
The study is open-label, expanded access study to provide continued OMS721 treatment for compassionate use to patients who have participated in clinical trial OMS721-TMA-001. Patients will be eligible if markers of disease activity, such as platelet count, LDH, and haptoglobin, were observed to improve during the study or if the patients disease activity remained stable, but they could be treated with a higher dose that may be beneficial. Safety measures of adverse events and laboratory measures will be monitored. Markers of disease activity, pharmacokinetics and ex vivo pharmacodynamics will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of thrombotic microangiopathy related to aHUS, TTP or stem cell transplant.
* Have completed treatment in clinical trial OMS721-TMA-001.
* Investigator determined that continued treatment with OMS721 could be beneficial.
* Aged 18 years or older.

Exclusion Criteria:

* Hypersensitivity to OMS721 or any excipients.
* Have a serious medical condition that increases the risk of OMS721 treatment to the patient.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michal Nowicki, MD, PhD, Principal Investigator — Medical University of Lodz